CLINICAL TRIAL: NCT04061070
Title: Effects of Trehalose and a Mix of Polyphenols on Endothelial Function, Oxidative Stress, Platelet Function and Autophagy in Vasculopathic Patients
Brief Title: Effects of Trehalose and Polyphenols in Vasculopathic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Peruzzi Mariangela (Unknown)
Responsible Party: Principal Investigator, Pasquale Pignatelli, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAD2307/2019 and 454/2020
Record Dates: First submitted 2019-07-24; First posted 2019-08-19 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2020-03

CONDITIONS: Oxidative Stress; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Dietary Supplements; Polyphenols

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention with the mix threalose plus polyphenols (Sham Comparator): The patients allocated in this arm will not treated with a mix of threalose plus polyphenols
  Interventions: Other: No Supplementation with mix of threalose plus polyphenols
- Intervention with the mix threalose plus polyhenols (Active Comparator): The patients allocated in this arm will treated with a mix of threalose plus polyphenols
  Interventions: Other: Supplementation with mix of threalose plus polyphenols

INTERVENTIONS:
Other: Supplementation with mix of threalose plus polyphenols — The patients will be treated with a mix of trehalose plus polyphenols for 60 days
  Arms: Intervention with the mix threalose plus polyhenols
Other: No Supplementation with mix of threalose plus polyphenols — The patients will not be treated with a mix trehalose plus polyphenols for 60 days
  Arms: No Intervention with the mix threalose plus polyphenols

SUMMARY:
Peripheral arterial disease (PAD) is an important manifestation of systemic atherosclerosis and is characterized by obstruction of the arteries of the lower extremities. PAD is usually associated with vascular complications that occur not only in peripheral circulation but also in cerebral and coronary trees (PubMed ID: 9892517). Endothelial dysfunction, reduced glucose oxidation, accumulation of toxic metabolites, alteration in nitric oxide (NO) generation and oxidative stress seem to play a role among the factors that contribute to reducing blood flow in PAD patients (PubMed ID: 17298965).

Hypertension is a risk factor for vascular disorders, including PAD. In fact, it has been shown that 55% of PAD patients are hypertensive. (PubMed ID: 15579058) PAD and hypertension patients have a risk of cardiovascular and cerebrovascular mortality increased two to three times compared to healthy subjects. The alteration of platelet function is implicated in the development and progression of atherosclerosis, as well as in the pathogenesis of acute cardiac ischemic events. Platelet activation is increased in patients with PAD and hypertension compared to healthy controls, suggesting a pro-thrombotic state.

Polyphenols are a class of natural, synthetic and semisynthetic substances with beneficial effects on human health. In particular, the polyphenols exert their beneficial effect through 1) the inhibition of NADPH oxidase (Nox2), which is crucial for the formation of reactive oxygen species (ROS); 2) an antiplatelet effects 3) the activation of autophagy. Trehalose is a natural disaccharide that performs multiple functions such as a protective action against oxidative stress, temperature changes, accumulation of protein aggregates and dehydration. Furthermore, recent evidence has shown that trehalose could prevent inflammatory responses induced by endotoxic shock both in vivo and in vitro.

Therefore the purpose of this work will be to determine in PAD and hypertension patients the effect of the intake of trehalose and a polyphenol mix on oxidative stress biomarkers, autophagic activity and endothelial dysfunction.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is an important manifestation of systemic atherosclerosis and is characterized by obstruction of the arteries of the lower limbs. PAD is usually associated with vascular complications that occur not only in peripheral circulation but also in cerebral and coronary trees (PubMed ID: 9892517). Intermittent claudication, the typical clinical manifestation of the disease that affects about a third of PAD patients, is identified by an alteration in blood flow to the lower extremities during exercise, worsens in 25% of patients and about 5% suffers an amputation (PubMed ID: 2647761). Arteries, arterioles, and capillaries that serve the skeletal muscle tissue distal to the site of the stenosis play a key role in the onset of claudication. Endothelial dysfunction, reduced glucose oxidation, accumulation of toxic metabolites, alteration in nitric oxide (NO) generation and oxidative stress seem to play a role among the factors that contribute to reducing blood flow in PAD patients (PubMed ID: 17298965). Nitric oxide (NO) is synthesized by L-arginine, is constitutively released by endothelial cells and serves to regulate vascular tone and to inhibit platelet function. NO is a potent anti-atherosclerotic molecule, as shown by an experimental study that shows that the integration of L-arginine reduces the progression of atherosclerosis. The generation of NO is reduced in patients with PAD and among the different mechanisms involved in the reduced generation of NO, the increase in oxidative stress could play a key role leading to accelerated degradation of NO or inhibition of NO synthase.

Increased serum levels of isoprostanes and autoantibodies against low-density oxidized lipoproteins confirm the increase in oxidative stress in these patients. Furthermore, the role of oxidative stress is confirmed by an intervention study in which PAD patients treated with propionyl-L-carnitine (6 g / day) for 7 days significantly increased the maximum distance traveled (MWD), an increase in bioavailability of NO and a reduction in oxidative stress.

The main risk factors involved in the onset of PAD include age, smoking, obesity, hyperlipemia and hypertension. Because hypertension is associated with the development of atherosclerosis, particularly in the coronary and cerebral circulation, it is also associated with an increased risk of developing PAD. In fact, of hypertensives at presentation, about 2-5% have intermittent claudication, with increasing prevalence with age. Otherwise, 35-55% of patients with PAD at presentation also show hypertension. Therefore, treatment of hypertension could lead to a reduction in the incidence of PAD. (PubMed ID:15579058) PAD patients have a risk of cardiovascular and cerebrovascular mortality increased two to three times compared to healthy subjects. The alteration of platelet function is implicated in the development and progression of atherosclerosis, as well as in the pathogenesis of acute cardiac ischemic events. Platelet activation is increased in patients with lower limb ischemia compared to healthy controls since it suggests a pro-thrombotic state.

Polyphenols are a class of natural, synthetic and semisynthetic molecules characterized by the presence of phenolic units. In recent decades, prospective and epidemiological studies that show potentially beneficial effects of these molecules on human health (for example on the cardiovascular and nervous systems). In particular, the polyphenols exert their beneficial effect through the inhibition of NADPH oxidase (Nox2), which is crucial for the formation of reactive oxygen species (ROS). There are several flavonoids that can exert antiplatelet effects for example by attenuating the process of platelet activation. Moreover, polyphenols can also exert beneficial effects through the activation of autophagy.

Autophagy is an intracellular cytoprotective process that mediates protein degradation, organelle turnover, and recycling of cytoplasmic components in conditions of nutrient deprivation and cellular stress (PubMed ID: 15068787). Furthermore, autophagy plays an important role in the removal of excess cellular ROS by maintaining a redox balance (PubMed ID: 27200146). The degraded materials in the autophagosome are then used for anabolic reactions, to sustain energy levels and provide simple molecules deriving from the degradation process that can be reused by cells for other functions. Autophagy, therefore, helps cells adapt to energy and stress changes by supporting cellular metabolism, homeostasis, and survival (PubMed ID: 18006683). The insufficient autophagic activity can contribute to cell death. Several studies have shown that inhibition of autophagic flow can contribute to the pathogenesis of cardiovascular diseases, diabetes, inflammatory disorders, cancer and physical stress (PubMed ID: 18191218).

Trehalose is a natural disaccharide composed of two glucose molecules linked by an α1-1-glycosidic bond, which is synthesized by lower organisms such as yeasts, insect bacteria, and plants but not by mammals. Trehalose performs multiple functions that distinguish it from other common disaccharides, including a protective action against various stressors, such as oxidative stress, temperature changes, accumulation of protein aggregates and dehydration (PubMed ID: 12626396). Furthermore, recent evidence has shown that trehalose could prevent inflammatory responses induced by endotoxic shock both in vivo and in vitro (PubMed ID: 17172986 and PubMed ID: 18555988). The oral administration of this disaccharide is able to drastically reduce the development and progression of neurodegenerative disorders, hepatic steatosis, renal damage, insulin resistance, atherosclerosis, post-ischemic cardiac remodelling and pancreatitis (PubMed ID: 22689910, PubMed ID: 21147367 and PubMed ID: 29724354) mainly through the stimulation of autophagy. Indeed, it has been shown that trehalose is a strong inducer of autophagy (PubMed ID: 17182613 ). Furthermore, our preliminary in vitro data showed that trehalose in combination with a mix of polyphenols (catechin and epicatechin) can reduce platelet activation, and oxidative stress and improves autophagic flow. Finally, we observed in the endothelial cells that the mix could increase the production of NO, angiogenetic property and cell viability.

ELIGIBILITY:
Inclusion Criteria for PAD patients (n=40):

1. claudication (defined as pain in the legs during walking which disappears within 10 minutes of standing);
2. ankle/brachial index (ABI), evaluated as an ankle/arm systolic blood pressure ratio using Doppler ultrasound on the worst resting leg;
3. stable condition without sudden changes in ABI (> 20%) in the last month before enrollment

Inclusion criteria for hypertensive patients (n=40):

Office systolic BP (SBP) values ≥140 mmHg and/or diastolic BP (DBP) values ≥90 mmHg (average of 3 repeated measurements made by the same doctor with an oscillometric automatic sphygmomanometer). Treatment with antihypertensive drugs, namely ACE inhibitors (ACEi), angiotensin receptor blockers (ARB), calcium channel blockers (CCB), thiazide/thiazide-like diuretics, loop diuretics, mineralocorticoid receptor antagonists (MRA), beta-blockers and alpha-blockers, were considered hypertensives.

Exclusion Criteria for PAD patients:

1. liver failure;
2. severe kidney disorders (serum creatinine [mt] 2.8 mg / dL);
3. acute cerebrovascular disease;
4. acute myocardial infarction;
5. smokers;
6. patients under treatment with antioxidants for at least 30 days before enrollment

Exclusion criteria for hypertensive patients:

Patients with diabetes mellitus or known history of ischemic heart disease, peripheral artery disease, and chronic renal failure were excluded.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change o oxidative stress biomarkers in PAD patients after mix supplementation of trehalose and polyphenols | 12 months
  Oxidative stress biomarkers such as Nox2 activity (pg/ml) production will be measured. Differences of these markers among patients taking or not the supplementation will be described.
Change o oxidative stress biomarkers in hypertensive patients after mix supplementation | 12 months
  To verify whether there is a reduction in the Nox2 activity in hypertensive patients after supplementation with the trehalose and polyphenols mix.

SECONDARY OUTCOMES:
Change of autophagy in PAD and hypertensive patients patients after mix supplementation of trehalose and polyphenols | 12 months
  Autophagy biomarkers such as LC3 (Arbitrary Unit) will be measured. Differences of this protein among patients taking or not the mix supplementation will be described. The relationship with oxidative stress markers will be described.
Change of endothelial function in PAD and hypertensive patients after mix supplementation of trehalose and polyphenols | 12 months
  To assess changes in endothelial function evaluated by Flow Mediated Dilation (FMD, %) analysis in patients taking or not the mix supplementation. The relationship with oxidative stress and autophagy will be described.
Change of systolic and diastolic pressure in PAD and hypertensive patients after mix supplementation of trehalose and polyphenols | 12 months
  To assess changes in systolic (mmHg) and diastolic (mmHg) pressure in patients taking or not the mix supplementation. The relationship with oxidative stress and autophagy will be described.
Analysis of maximal walking distance (MWD) in PAD patients after mix supplementation of trehalose and polyphenols | 12 months
  To assess changes in MWD (meters) evaluated by treadmill test in patients taking or not the mix supplementation. The relationship with oxidative stress, autophagy and endothelial function will be described.
Analysis of maximal walking time (MWT) in PAD | 12 months
  o assess changes in MWD (seconds) evaluated by treadmill test in patients taking or not the mix supplementation. The relationship with oxidative stress, autophagy and endothelial function will be described.
Analysis of blood pressure in hypertensive patients after mix supplementation of trehalose and polyphenols | 12 months
  o assess changes in blood pressure in patients taking or not the mix supplementation. The relationship with oxidative stress, autophagy and endothelial function will be described.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Umberto I Policlinico di Roma, Sapienza Università di Roma, Roma, Italia
  - Umberto I Policlinico di Roma, Sapienza Università di Roma, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Criqui MH, Denenberg JO. The generalized nature of atherosclerosis: how peripheral arterial disease may predict adverse events from coronary artery disease. Vasc Med. 1998;3(3):241-5. doi: 10.1177/1358836X9800300311. PMID 9892517
- [Result] Loffredo L, Marcoccia A, Pignatelli P, Andreozzi P, Borgia MC, Cangemi R, Chiarotti F, Violi F. Oxidative-stress-mediated arterial dysfunction in patients with peripheral arterial disease. Eur Heart J. 2007 Mar;28(5):608-12. doi: 10.1093/eurheartj/ehl533. Epub 2007 Feb 13. PMID 17298965
- [Result] Dormandy J, Mahir M, Ascady G, Balsano F, De Leeuw P, Blombery P, Bousser MG, Clement D, Coffman J, Deutshinoff A, et al. Fate of the patient with chronic leg ischaemia. A review article. J Cardiovasc Surg (Torino). 1989 Jan-Feb;30(1):50-7. PMID 2647761
- [Result] Levine B, Klionsky DJ. Development by self-digestion: molecular mechanisms and biological functions of autophagy. Dev Cell. 2004 Apr;6(4):463-77. doi: 10.1016/s1534-5807(04)00099-1. PMID 15068787
- [Result] Li F, Lang F, Zhang H, Xu L, Wang Y, Hao E. Role of TFEB Mediated Autophagy, Oxidative Stress, Inflammation, and Cell Death in Endotoxin Induced Myocardial Toxicity of Young and Aged Mice. Oxid Med Cell Longev. 2016;2016:5380319. doi: 10.1155/2016/5380319. Epub 2016 Apr 21. PMID 27200146
- [Result] Mizushima N. Autophagy: process and function. Genes Dev. 2007 Nov 15;21(22):2861-73. doi: 10.1101/gad.1599207. PMID 18006683
- [Result] Levine B, Kroemer G. Autophagy in the pathogenesis of disease. Cell. 2008 Jan 11;132(1):27-42. doi: 10.1016/j.cell.2007.12.018. PMID 18191218
- [Result] Elbein AD, Pan YT, Pastuszak I, Carroll D. New insights on trehalose: a multifunctional molecule. Glycobiology. 2003 Apr;13(4):17R-27R. doi: 10.1093/glycob/cwg047. Epub 2003 Jan 22. PMID 12626396
- [Result] Minutoli L, Altavilla D, Bitto A, Polito F, Bellocco E, Lagana G, Giuliani D, Fiumara T, Magazu S, Ruggeri P, Guarini S, Squadrito F. The disaccharide trehalose inhibits proinflammatory phenotype activation in macrophages and prevents mortality in experimental septic shock. Shock. 2007 Jan;27(1):91-6. doi: 10.1097/01.shk.0000235092.76292.bc. PMID 17172986
- [Result] Minutoli L, Altavilla D, Bitto A, Polito F, Bellocco E, Lagana G, Fiumara T, Magazu S, Migliardo F, Venuti FS, Squadrito F. Retracted: Trehalose: a biophysics approach to modulate the inflammatory response during endotoxic shock. Eur J Pharmacol. 2008 Jul 28;589(1-3):272-80. doi: 10.1016/j.ejphar.2008.04.005. Epub 2008 Apr 12. PMID 18555988
- [Result] Schaeffer V, Lavenir I, Ozcelik S, Tolnay M, Winkler DT, Goedert M. Stimulation of autophagy reduces neurodegeneration in a mouse model of human tauopathy. Brain. 2012 Jul;135(Pt 7):2169-77. doi: 10.1093/brain/aws143. Epub 2012 Jun 10. PMID 22689910
- [Result] Arai C, Arai N, Mizote A, Kohno K, Iwaki K, Hanaya T, Arai S, Ushio S, Fukuda S. Trehalose prevents adipocyte hypertrophy and mitigates insulin resistance. Nutr Res. 2010 Dec;30(12):840-8. doi: 10.1016/j.nutres.2010.10.009. PMID 21147367
- [Result] Sciarretta S, Yee D, Nagarajan N, Bianchi F, Saito T, Valenti V, Tong M, Del Re DP, Vecchione C, Schirone L, Forte M, Rubattu S, Shirakabe A, Boppana VS, Volpe M, Frati G, Zhai P, Sadoshima J. Trehalose-Induced Activation of Autophagy Improves Cardiac Remodeling After Myocardial Infarction. J Am Coll Cardiol. 2018 May 8;71(18):1999-2010. doi: 10.1016/j.jacc.2018.02.066. PMID 29724354
- [Result] Sarkar S, Davies JE, Huang Z, Tunnacliffe A, Rubinsztein DC. Trehalose, a novel mTOR-independent autophagy enhancer, accelerates the clearance of mutant huntingtin and alpha-synuclein. J Biol Chem. 2007 Feb 23;282(8):5641-52. doi: 10.1074/jbc.M609532200. Epub 2006 Dec 20. PMID 17182613
- [Result] Clement DL, De Buyzere ML, Duprez DA. Hypertension in peripheral arterial disease. Curr Pharm Des. 2004;10(29):3615-20. doi: 10.2174/1381612043382819. PMID 15579058
- [Derived] Martinelli O, Peruzzi M, Bartimoccia S, D'Amico A, Marchitti S, Rubattu S, Chiariello GA, D'Ambrosio L, Schiavon S, Miraldi F, Saade W, D'Abramo M, Pingitore A, Loffredo L, Nocella C, Forte M, Pignatelli P. Natural Activators of Autophagy Increase Maximal Walking Distance and Reduce Oxidative Stress in Patients with Peripheral Artery Disease: A Pilot Study. Antioxidants (Basel). 2022 Sep 18;11(9):1836. doi: 10.3390/antiox11091836. PMID 36139910